CLINICAL TRIAL: NCT01101464
Title: A Single-center, Open-label, 2-way Crossover Relative Bioavailability and Safety Trial With Two Differing Strength Tablets (3 x 5 mg vs. 1 x 15 mg) of Sublingually Administered Org 5222 in Subjects With Schizophrenia or Schizoaffective Disorder.
Brief Title: A Trial to Determine Whether Two Differing Strength Tablets (3 x 5 mg Versus 1 x 15 mg) of Sublingually Org 5222 (Asenapine) Are Safe and Equal in Subjects With Schizophrenia or Schizoaffective Disorder (P05937)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: P05937
Record Dates: First submitted 2010-03-03; First posted 2010-04-12 (Estimated); Results first posted 2010-10-13 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — asenapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Asenapine Sequence 1 (Experimental)
  Interventions: Drug: Asenapine 3x5mg followed by 1x15mg
- Asenapine Sequence 2 (Experimental)
  Interventions: Drug: Asenapine 1x15mg followed by 3x5mg

INTERVENTIONS:
Drug: Asenapine 3x5mg followed by 1x15mg — Three 5 mg sublingual tablets (15 mg) given twice daily for 2 days followed by one 15 mg sublingual tablet given twice daily for 1.5 days
  Other Names: Org 5222, SCH 900274
  Arms: Asenapine Sequence 1
Drug: Asenapine 1x15mg followed by 3x5mg — One 15 mg sublingual tablet given twice daily for 2 days followed by three 5 mg sublingual tablets (15 mg) given twice daily for 1.5 days.
  Arms: Asenapine Sequence 2

SUMMARY:
A trial to compare if one 15 mg under the tongue tablet is equal to three 5 mg under the tongue tablets of Org 5222 (asenapine) in subjects with schizophrenia or schizoaffective disorder delivered.

ELIGIBILITY:
Inclusion Criteria:

* must provide written informed consent after the scope and nature of the investigation has been explained to them, but before signing any trial-related activities, including screening evaluations;
* must be at least 18 and less than 65 years of age;
* can be either male or female; females must be either surgically sterile, postmenopausal for at least 1 year, or non-pregnant using a method of birth control that was acceptable to the investigator;
* must be able to speak, read and understand English and be able to respond to questions and follow simple instructions;
* must be diagnosed at the screening interview according to Diagnostic & Statistical Manual of Mental Disorders, 4th edition (DSM-IV), with non-first episode schizophrenia or schizoaffective disorder (295.70); if schizophrenia, must be of the following types: schizophrenia of the paranoid type (295.30), schizophrenia of the disorganized type (295.10), schizophrenia of the catatonic type (295.20), schizophrenia of the undifferentiated type (295.90), schizophrenia of the residual type (295.60);
* must have discontinued all use of all antipsychotic medication except depot neuroleptics at least 3 days prior to baseline. For depot neuroleptics, subjects must have completed 1 dosing interval by the baseline interview;
* must not have taken any experimental medication for at least 30 days prior to baseline;
* with hypothyroidism, diabetes, high blood pressure, or chronic respiratory conditions can be considered as candidates for enrollment in the trial if their conditions are stable, they are receiving standard therapies for the condition, the prescribed dose and regimen of medication is stable for at least 3 months, and all appropriate clinical and laboratory parameters are within the clinically acceptable limits for the condition, and
* must be willing to remain in the hospital a minimum of 14 days to approximately 17 days (minimum of a 3- to a maximum of a 7-day washout period, a minimum of an 8-day in-patient period, and a possible 3-day stabilization period, if needed, prior to discharge).

Exclusion Criteria:

* they have any untreated or uncompensated clinically significant renal, endocrine, hepatic, respiratory, cardiovascular, hematologic, immunologic, or cerebrovascular disease, or malignancy;
* they are considered obese by the investigator (e.g., greater than 30% above ideal body weight);
* they have a seizure disorder or are taking anticonvulsants to prevent seizures;
* they have any clinically relevant electrocardiogram (ECG) abnormalities at the screening visit (Day -2) or at baseline (Day 0);
* they have a history of a clinically significant cardiac event that required resuscitation;
* at the screening visit, on admission to the trial, during the washout period or at baseline (Day 0), they have any clinically significant abnormal laboratory, vital sign, or physical examination findings which, in the opinion of the investigator, would preclude trial participation;
* they require concomitant treatment with hypnotics (for sleep induction) other than chloral hydrate ≤3000 mg/day, or Ambien (zolpidem tartrate) ≤10 mg qhs, and (for agitation) a benzodiazepine such as lorazepam, ≤10 mg/day;
* they have a score greater than mild at baseline (score >2) on any item of the Abnormal Involuntary Movement Scale (AIMS) assessment at screening and/or require ongoing treatment with anticholinergic medication beyond baseline (Day 0);
* they have a history of significant drug and/or alcohol abuse (according to DSM-IV criteria 305.00) within 30 days before the screening visit;
* they have a confirmed positive result on the alcohol/drug screen test for alcohol, illegal (excluding marijuana), or non-prescribed drugs at screening or at hospital admission;
* they had a primary psychiatric diagnosis (according to DSM-IV criteria) other than schizophrenia or schizoaffective disorder;
* they are actively suicidal at the screening visit, or become so at admission to the hospital, during the washout period, or at baseline (Day 0);
* they have a Clinical Global Impression (CGI) (Severity of Illness) rating greater than moderately ill (score >4) at screening or baseline;
* they are non-compliant (>25%) during the washout period (including baseline Day 0); or,
* they are pregnant, intend to become pregnant during the course of the trial, or are currently nursing mothers during the course of the trial.
* require concomitant medications that are substrates, inhibitors, or inducers of Cytochrome P450 CYP3A4.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2002-10; Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All subjects rec'd asenapine 5mg BID on Day 1 & 10mg BID on Day 2. Subjects rec'd 15mg BID (either 3x5mg or 1x15mg according to their randomized sequence) from the morning dose on Day 3 through the morning dose on Day 5, followed by the alternate treatment (either 3x5mg or 1x15mg) from the evening dose on Day 5 through the morning dose on Day 7.
Groups:
- Asenapine, (3) 5mg Then (1) 15 mg: Three 5 mg sublingual tablets (15 mg) given twice daily for 2 days followed by one 15 mg sublingual tablet given twice daily for 1.5 days.
- Asenapine, (1) 15 mg Then (3) 5 mg: One 15 mg sublingual tablet given twice daily for 2 days followed by three 5 mg sublingual tablets (15 mg) given twice daily for 1.5 days.
Period: Day 1 Through AM Dose of Day 5
Arm/Group | Asenapine, (3) 5mg Then (1) 15 mg | Asenapine, (1) 15 mg Then (3) 5 mg
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0
Period: PM Dose of Day 5 Through AM Dose of Day7
Arm/Group | Asenapine, (3) 5mg Then (1) 15 mg | Asenapine, (1) 15 mg Then (3) 5 mg
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Asenapine, (3) 5 mg Then (1) 15 mg: Three 5 mg sublingual tablets (15 mg) given twice daily for 2 days followed by one 15 mg sublingual tablet given twice daily for 1.5 days
- Total: Total of all reporting groups
Arm/Group | Asenapine, (3) 5 mg Then (1) 15 mg | Asenapine, (1) 15 mg Then (3) 5 mg | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic Parameter of Maximum Plasma Concentration (Cmax) of Two Differing Tablet Strengths (3 x 5 mg and 1 x 15 mg) of Sublingually Administered Org 5222 (Asenapine)
Description: The primary objective is to compare the bioavailability using pharmacokinetic parameter of maximum plasma concentration (Cmax) of two differing tablet strengths (3 x 5 mg and 1 x 15 mg) of sublingually administered Org 5222
  Measurements were performed after each cross-over period: Day 5 measurement for 3x5mg for participants from Sequence 1 and 1x15mg for participants from Sequence 2; Day 7 measurement for 1x15mg for participants from Sequence 1 and 3x5mg for participants from Sequence 2.
Time Frame: Day 5 & Day 7
Population: All participants were included in both treatment comparisons (as per cross over design).
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Asenapine 3x5mg: Three 5 mg sublingual tablets (15 mg) given twice daily for 2 or 1.5 days (depending on sequence of participant)
- Asenapine 1x15mg: One 15 mg sublingual tablet given twice daily for 2 or 1.5 days (depending on sequence of participant)
Arm/Group | Asenapine 3x5mg | Asenapine 1x15mg
Number analyzed (Participants) | 8 | 8
ng/mL | 6.89 (3.08) | 6.38 (2.76)

2. Primary Outcome: Pharmacokinetic Parameter of Time of Occurrence of Cmax (Tmax) of Two Differing Tablet Strengths (3 x 5 mg and 1 x 15 mg) of Sublingually Administered Org 5222 (Asenapine)
Description: The primary objective is to compare the bioavailability using pharmacokinetic parameter of time of occurrence of Cmax (Tmax) of two differing tablet strengths (3 x 5 mg and 1 x 15 mg) of sublingually administered Org 5222.
  Measurements were performed after each cross-over period: Day 5 measurement for 3x5mg for participants from Sequence 1 and 1x15mg for participants from Sequence 2; Day 7 measurement for 1x15mg for participants from Sequence 1 and 3x5mg for participants from Sequence 2
Time Frame: Day 5 & Day 7
Population: All participants were included in both treatment comparisons (as per cross over design).
Measure: Mean (Full Range); unit: Hours
Arm/Group | Asenapine 3x5mg | Asenapine 1x15mg
Number analyzed (Participants) | 8 | 8
Hours | 1.25 [0.5 to 2.0] | 1.00 [0.5 to 3.0]

3. Primary Outcome: Pharmacokinetic Parameter of Area Under the Curve (AUC) of Two Differing Tablet Strengths (3 x 5 mg and 1 x 15 mg) of Sublingually Administered Org 5222 (Asenapine)
Description: The primary objective is to compare the bioavailability using pharmacokinetic parameter of area under the curve (AUC) of two differing tablet strengths (3 x 5 mg and 1 x 15 mg) of sublingually administered Org 5222.
  Measurements were performed after each cross-over period: Day 5 measurement for 3x5mg for participants from Sequence 1 and 1x15mg for participants from Sequence 2; Day 7 measurement for 1x15mg for participants from Sequence 1 and 3x5mg for participants from Sequence 2.
Time Frame: Day 5 & Day 7
Population: All participants were included in both treatment comparisons (as per cross over design).
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Asenapine 3x5mg | Asenapine 1x15mg
Number analyzed (Participants) | 8 | 8
ng*h/mL | 41.3 (18.2) | 41.1 (17.1)

ADVERSE EVENTS:
Description: All subjects rec'd asenapine 5mg BID on Day 1 & 10mg BID on Day 2. Subjects rec'd 15mg BID (either 3x5mg or 1x15mg according to their randomized sequence) from the morning dose on Day 3 through the morning dose on Day 5, followed by the alternate treatment (either 3x5mg or 1x15mg) from the evening dose on Day 5 through the morning dose on Day 7.
Arm/Group | Asenapine, (3) 5 mg Then (1) 15 mg | Asenapine, (1) 15 mg Then (3) 5 mg
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 2/4 | 3/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asenapine, (3) 5 mg Then (1) 15 mg (N=4) | Asenapine, (1) 15 mg Then (3) 5 mg (N=4)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Extrapyramidal disosrder (Nervous system disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All publications must be based on data validated by Organon. Any such communication will first be submitted to Organon, at least 6 weeks ahead of time for written consent. Organon shall have the right to make its consent conditional upon proper representation of the interpretation of both Organon and the investigator. In any communication concerning this trial, the authors of this protocol will be included in the list of authors.